CLINICAL TRIAL: NCT01869842
Title: Randomized Controlled Study of the Traditional Percutaneous Coronary Intervention and Intervention Using Optical Coherence Tomography of Incomplete Stent Adhesion and Extent of the Formation of Neointima by Resolute Zotarolimus-eluting Stent Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2011-0070
Record Dates: First submitted 2013-05-31; First posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease; Stable Angina; Unstable Angina
Keywords: Resolute zotarolumus-eluting stent; optical coherence tomography
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- DM, angio group (Active Comparator)
  Interventions: Procedure: percutaneous coronary intervention
- DM, OCT group (Experimental)
  Interventions: Procedure: OCT-guided percutaneous coronary intervention
- non DM, angio group (Active Comparator)
  Interventions: Procedure: percutaneous coronary intervention
- non DM, OCT group (Experimental)
  Interventions: Procedure: OCT-guided percutaneous coronary intervention

INTERVENTIONS:
Procedure: percutaneous coronary intervention — the traditional percutaneous coronary intervention by Resolute zotarolimus-eluting stent insertion
  Arms: DM, angio group
Procedure: OCT-guided percutaneous coronary intervention — the percutaneous coronary intervention using optical coherence tomography by Resolute zotarolimus-eluting stent insertion
  Arms: DM, OCT group
Procedure: percutaneous coronary intervention — the traditional percutaneous coronary intervention by Resolute zotarolimus-eluting stent insertion
  Arms: non DM, angio group
Procedure: OCT-guided percutaneous coronary intervention — the percutaneous coronary intervention using optical coherence tomography by Resolute zotarolimus-eluting stent insertion
  Arms: non DM, OCT group

SUMMARY:
Optical coherence tomography (OCT) after the stent procedure to improve the adhesion and expansion, or incomplete uncovered struts attached to the main track. OCT in clinical areas by improving the parameters of the best stent will be useful. However, for better results for optical coherence tomography in percutaneous interventions have little useful data on the role. Randomized controlled study of the traditional percutaneous coronary intervention and intervention using optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

* Single lesion in a Single vessel
* Reference vessel diameter 2.5 - 3.5 mm
* Lesion length ≤ 34 mm and ≤ 34 mm stent length
* Stable angina requiring revascularization, patients with unstable angina
* The patient has no difficulty to enforce the follow-up angiography
* Patient is ≥ 20 years old

Exclusion Criteria:

* Lesions with graft vessel, thrombosis, restenosis, and bifurcation requiring 2 stents
* Reference vessel diameter < 2.5 mm or > 4.0mm
* Contraindication to anti-platelet agents
* Treated with any DES within 3 months at other vessel
* Creatinine level ≥ 2.0 mg/dL or ESRD
* Severe hepatic dysfunction (3 times normal reference values)
* Patients with LVEF < 30%
* Life expectancy 1 year
* Lesions with CTO or left main
* Target vessel of ST-elevation MI
* Lesions requiring overlapped stenting or more than 2 DES in each vessel
* Heavy calcified lesions (definite calcified lesions on angiogram)
* Far distal or tortuous lesions having difficulties in OCT evaluation or follow-up OCT
* Pregnant women or women with potential childbearing

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ratio of the stent strut | Angiographic follow-up with OCT at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea